CLINICAL TRIAL: NCT07107217
Title: Camrelizumab in Combination With Chemotherapy as Neoadjuvant Treatment in Patients With Early or Locally Advanced Triple-negative Breast Cancer
Acronym: Camella
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 15.07.2025
Record Dates: First submitted 2025-07-17; First posted 2025-08-06 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Early Breast Cancer; Neoadjuvant Therapy; Camrelizumab
MeSH Terms: conditions — Breast Neoplasms | interventions — camrelizumab; CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neadjuvant chemotherapy (Experimental): 4 course ddAC (doxorubicin 60 mg/m² as an and cyclophosphamide 600 mg/m² on day 1 every 2 weeks + filgrastim (G-CSF) subcutaneously on days 2-6 ) + paclitaxel 80 mg/m² + carboplatin AUC2 on day 1 every 1 weeks a total of 12 weeks with camrelizumab at a dose of 200 mg once every 2 weeks for a total of 20 weeks.
  Interventions: Drug: Camrelizumab; Drug: Doxorubicin +cyclophosphamide+ filgrastimum; Drug: carboplatin + paclitaxel (CP)

INTERVENTIONS:
Drug: Camrelizumab — 200 mg by intravenous (iv.) infusion every 2 weeks (Q2W) for 10 times
Drug: Doxorubicin +cyclophosphamide+ filgrastimum — Doxorubicin 60mg/m² + cyclophosphamide 600 mg/m² on Day 1 of Cycles 1-4 (Q2W) of the first neoadjuvant phase of the study, IV infusion. filgrastim (G-CSF) subcutaneously on days 2-6 of Cycles 1-4
Drug: carboplatin + paclitaxel (CP) — carboplatin AUC 2 and paclitacel 80 mg/m² will be given on day 1 every 12 weeks of the second neoadjuvant phase of the study, IV infusion.

SUMMARY:
To explore the application of Camrelizumab with chemotherapy as neoadjuvant treatment of early-stage TNBC. Phase II clinical study of Camrelizumab in neoadjuvant treatment of early-stage TNBC is proposed. The study aims to evaluate the efficacy and safety of Camrelizumab and to provide a new treatment option for neoadjuvant treatment of early-stage TNBC.

DETAILED DESCRIPTION:
This study is a single center, non blinded, randomized phase II clinical trial. A total of 40 patients early-stage T3-4NanyM0 any TanyN+M0 TNBC, who meet the inclusion and exclusion criteria, are planned to be enrolled.

Patients will receive neoadjuvant chemotherapy as 4 course ddAC (doxorubicin 60 mg/m² as an and cyclophosphamide 600 mg/m² on day 1 every 2 weeks) + paclitaxel 80 mg/m² + carboplatin AUC2 on day 1 every 1 weeks a total of 12 weeks with camrelizumab at a dose of 200 mg once every 2 weeks for a total of 16 weeks.

Imaging assessments will be conducted every 4 weeks during the neoadjuvant treatment phase. After the neoadjuvant treatment is completed, surgery will be performed within 4 weeks of the last study drug administration. Whether to receive adjuvant treatment after surgery will be determined by the investigator. The primary endpoint of the study is the pathological complete response (pCR) rate. Secondary endpoints include objective response rate (ORR), event-free survival (EFS), overall survival (OS), and safety. During the follow-up phase, survival follow-up will be conducted every 3 months (±28 days) in the first year and every 6 months (±28 days) thereafter, until disease progression, disease recurrence, or until 3 years after the last patient is enrolled (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

1) 18-65 Years, female; 2) Histologically documented Triple Negative Breast Cancer (TNBC) patients; 3) Previously untreated non-metastatic (M0) TNBC, T3-4NanyM0 или TanyN+M0 3) Promising radical surgical treatment; 4) At least one measurable lesion according to RECIST 1.1; 5) Life expectancy is not less than 3 months; 6) ECOG: 0～1; 7) Adequate function of major organs meets the following requirements:

8) Neutrophils ≥ 1.5×10^9/L Hemoglobin ≥ 90g/L Platelets ≥ 100×10^9/L Total bilirubin≤ 1.5 × the upper limit of normal (ULN) ALT and AST ≤ 2.5 × ULN Serum creatinine ≤1.5 × ULN, Endogenous creatinine clearance ≥50mL/min;

9) Left ventricular ejection fraction (LVEF) ≥50% or ≥ limit of normal (LLN) was evaluated by echocardiography (ECHO) or Multigated Acquisition (MUGA); 10) Women with childbearing potential who are must agree to take effective contraceptive measures during the study period and ≥120 days after the last administration of the study drug, and must have a negative serum pregnancy test result within 7 days prior to initiation of study drug.

11) The patient voluntarily joined the study, signed an informed consent form, had good compliance, and cooperated with follow-up;

Exclusion Criteria:

1. Has participated in an interventional clinical study with an investigational compound within 4 weeks prior to initiation of study treatment;
2. Prior treatment with anti-cytotoxic T-lymphocyte-associated protein 4 (anti-CTLA-4), anti-programmed death-1 (anti-PD-1), and anti-PD-L1 therapeutic antibodies;
3. Has a history of invasive malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer;
4. Active or history of autoimmune disease or immune deficiency diseases except history of autoimmune-related hypothyroidism, controlled Type 1 diabetes mellitus;;
5. Has a history of (non-infectious) pneumonitis, interstitial lung disease or uncontrollable systematicness diseases, including pulmonary fibrosis, acute lung disease, etc.;
6. Administration of a live attenuated vaccine within 30 days prior to initiation of study treatment or anticipation of need for such a vaccine during the study;
7. Has active infection (CTCAE≥2) needed the treatment of antibiotic within 2 weeks prior to initiation of study treatment;
8. Has a history of serious cardiovascular disease, including myocardial infarction, acute coronary syndrome or coronary angioplasty/stent implantation/bypass grafting history in the past 6 months, and have level II-IV congestion Heart failure (CHF), or III NYHA and IV CHF history;
9. Prior allogeneic stem cell or solid organ transplantation
10. History of neurological or psychiatric disorders, including schizophrenia, severe depressive disorder, bipolar disorder, etc.;
11. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first administration of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
12. History of severe hypersensitivity reactions to other monoclonal antibodies, or intravenous infusion, or Doxorubicin, or cyclophosphamide, or paclitaxel, or carboplatine
13. Female patients during pregnancy and lactation, fertile women with positive baseline pregnancy tests or women of childbearing age who are unwilling to take effective contraceptive measures throughout the trial;
14. Any other situation evaluated by researchers.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) | The outcome was changed from 19 weeks at the time of results entry as the treatment period was actually 20 weeks and the outcome was assessed 4-6 weeks after treatment when surgery took place.
  Pathologic response will be assessed in the surgically resected cancer and lymph nodes after completion of all chemotherapy by the local pathologist as part of routine care. Pathologic complete response is defined as no invasive cancer in the resected breast tissue and lymph nodes (ypT0/Tis, ypN0).

SECONDARY OUTCOMES:
objective response rate (ORR) | average 18 months
Disease-free Survival | expected average 48 months
  Defined as the time between Day 1 Cycle 1 to breast cancer progression
Overall Survival | approximately 48 months
  Defined as the time between Day 1 Cycle 1 to date of death from any cause

IPD SHARING:
Plan to Share IPD: No